CLINICAL TRIAL: NCT03501056
Title: Phase II Randomized Comparison Clinical Trial of Target Activated CIK for Advanced Lung Cancer
Brief Title: Study of Activated Cytokine-induced Killer Armed With Bispecific Antibody for Advanced Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Benhealth Biopharmaceutical (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD3-MUC1 in lung cancer
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05

CONDITIONS: Advanced Lung Cancer
Keywords: PD-1 activated CIK; MUC1; Bispecific antibody; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: This is a phase II clinical trial of single-center, and it will divide into three groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the method of minimum randomized dynamic random by the interactive network response system (IWRS),Participants were assigned to three groups,receive cryotherapy,conventional therapy, and activated CIK armed with anti-CD3-MUC1 bispecific antibody together with cryotherapy .every participant has a unique identification number and emergency letter which have the information of group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cryotherapy (Experimental): the maximum tumor length≥2 cm，cool down the lesion,result in degeneration, necrosis or loss of the lesion.
  Interventions: Procedure: Cryotherapy
- Cryotherapy & Activated CIK and bispecific antibody (Active Comparator): the maximum tumor length≥2cm, use cryotherapy. the maximum tumor length<2 cm,Biological/Vaccine:Activated CIK and bispecific antibody CIK cells was activated by PD-1 inhibitor and bispecific antibody of anti-CD3/MUC1
  Interventions: Biological: Activated CIK and CD3-MUC1 Bispecific Antibody in Treating Lung cancer; Procedure: Cryotherapy
- conventional therapy (No Intervention): In this group, the patients will receive no special treatment and as a control group. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).

INTERVENTIONS:
Biological: Activated CIK and CD3-MUC1 Bispecific Antibody in Treating Lung cancer — CIK cells was activated by PD-1 inhibitor and bispecific antibody of anti-CD3/MUC1
  Arms: Cryotherapy & Activated CIK and bispecific antibody
Procedure: Cryotherapy — the maximum tumor length≥2 cm，cool down the lesion,result in degeneration, necrosis or loss of the lesion.
  Arms: Cryotherapy & Activated CIK and bispecific antibody; cryotherapy

SUMMARY:
This is a phase II Randomized comparison clinical trial of activated CIK armed with anti-CD3-MUC1 bispecific antibody for advanced lung cancer. And the aim of this research is to study the clinical efficacy and safety of activated CIK armed with anti-CD3-MUC1 bispecific antibody for lung cancer.

DETAILED DESCRIPTION:
Primary pulmonary carcinoma is one of the most common malignancies in China, ranking first in all malignant tumors and mortality.Immunetherapy is considered to be one of the most promising means of human against cancer. This is a phase II clinical trial of single- center, The investigators plan to recruit for 90 patients with advanced lung cancer,and all patients are divided into three groups.one group will receive cryotherapy, one group will receive conventional therapy，and the rest one will receive mixed liquor of activated CIK and anti-CD3-MUC1 bispecific antibody together with cryotherapy.

The result of this study was statistic and analysed with the record of Response Evaluation Criteria In Solid Tumors(RECIST1.1) evaluation standard.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* The patient is diagnosed as advanced lung cancer,MUC1 is positive
* There is at least one tumor should be measured,and length≥10mm of focus not at lymph node or length≥10mm of focus at lymph node
* The patient can't tolerate system(systemic chemotherapy/molecular targeted therapy) or local therapies
* If the patient received adjuvant chemotherapy after local treatment,the time should be more than 4 weeks after the end of chemotherapy, and disease progression or metastasis patients can also assigned into the group
* The time of surgical treatment≥ 3 months ;At the end of the intervention,radiotherapy and the end of the ablation time is more than 4 weeks
* The expected survival time ≥12 weeks
* The patient did not took any antitumor drugs within 4 weeks(any antitumor drugs, Chinese patent medicine including Delisheng injection,Kanglaite injection, Aidi injection
* No serious disease are conflicts with the solution(such as autoimmune disease,immunodeficiency,organ transplantation)
* Sign the informed consent

Exclusion Criteria:

* medium or above ascites
* Patient of second primary tumor or multiple primary cancer
* Patients of T cell lymphoma、myeloma,and patients are using immunosuppressant
* Systemic autoimmune diseases, allergic constitution or immunocompromised patients
* Patients of chronic diseases need immune stimulant or hormone therapy
* Patients of active bleeding or coagulant function abnormality（PT>16s、APTT>43s、TT>21s、INR≥2）,and patients of bleeding tendency or are receiving thrombolysis and anticoagulation and antiplatelet therapy
* Women who is pregnant or during breast feeding or plan to pregnant in 2 years,and not willing to contraception during the test
* Patients with brain、dura mater metastases or history of psychogenic
* Gastrointestinal bleeding in the past six months or have clear gastrointestinal bleeding tendency,such as: patients of local active ulcerative lesions, defecate occult blood + + above shall not enter into group; defecate occult blood + depend on gastroscopy
* Patients with severe stomach/esophageal varices and need for intervention treatment
* Patients with abdominal fistula, gastrointestinal perforation or abdominal abscess within 4 weeks before the first treatment
* Positive for HIV antibody
* Patients who are allergic to computed tomography (CT) and magnetic resonance imaging (MRI) contrast agents at the same time, can't imaging assay
* Patients accepted any experimental drugs or pilot medical apparatus and instruments in the past 4 weeks of first treatment
* Other reasons the researchers think not suitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  ORR.The proportion of patients who had a best response rating of complete response and partial response.

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  PFS.The time of patients from randomization to death caused by the progression of the tumor or any cause.
Time tumor progression | 1 year
  TTP.The time of patient from randomization to objective progress of the tumor.
Disease control rate | 1 year
  DCR.The proportion of patients who had a best response rating of complete response, partial response,or stable disease.
Overall survival | 3 years
  OS.The time of patient from randomization to death caused by any cause
Symptom remission rate | 1 year
  SRR. The proportion of symptoms are alleviated in all evaluative cases.

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, Doctor, Study Chair — Guangzhou Fuda Cancer Hospital
Locations (1):
- Institutional Review Board of Guangzhou Fuda Cancer Hospital, Guangzhou, Guangdong, China